CLINICAL TRIAL: NCT06602180
Title: Scapular Proprioceptive Neuromuscular Facilitation and Activity Oriented Antiedema Proprioceptive Therapy on Shoulder Dysfunction Post Matectomy Lymphedema
Brief Title: Scapular PNF and Activity Oriented Antiedema Proprioceptive Therapy on Shoulder Dysfunction Post Matectomy Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Abdalfattah Ahmed Selim, Master of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 152427
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Upper Limb Edema
MeSH Terms: interventions — tapasin; Methods; carbohydrate-deficient transferrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double : participant ,investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exprimental group A (Experimental): Thirty-one patients will receive: Scapular PNF technique, (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (CDT).
  Interventions: Other: Scapular PNF technique, (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT).
- Experimental: group B (Experimental): Thirty-one patients will receive Scapular PNF technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT))
  Interventions: Other: Scapular PNF technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT))
- Experimental: group C: (Experimental): Thirty-one patients will receive Activity-Oriented Antiedema Proprioceptive Therapy (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT)
  Interventions: Other: Activity-Oriented Antiedema Proprioceptive Therapy (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT)

INTERVENTIONS:
Other: Scapular PNF technique, (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT). — Complex or combined decongestive physical therapy (CDT):
  skin care and patient education, manual lymphatic drainage MLD, joints exercises, and compression garments.
  Scapular PNF:
  Proprioceptive Neuromuscular Facilitation (PNF) is treatment approach that focus on motor learning, helps the patient to relax, improves coordination, and normalizes the motion. The repeated contractions technique increases active range of motion and strength and guides the patient's motion towards the desired motion,
  TAPA involves an intervention protocol composed of:
  10-min neuro dynamics oriented to the activity 10-min proprioceptive neuromuscular facilitation activities. 10-min proprioceptive anti-edema bandaging, including patient and/or caretaker instructions for placement, as well as assistance on techniques to use for performing everyday activities,
  Arms: Exprimental group A
Other: Scapular PNF technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT)) — Proprioceptive Neuromuscular Facilitation (PNF) is treatment approach that focus on motor learning, helps the patient to relax, improves coordination, and normalizes the motion. The repeated contractions technique increases active range of motion and strength and guides the patient's motion towards the desired motion,
  Complex or combined decongestive physical therapy (CDT):
  skin care and patient education, manual lymphatic drainage MLD, joints exercises, and compression garments
  Arms: Experimental: group B
Other: Activity-Oriented Antiedema Proprioceptive Therapy (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT) — Activity-Oriented Proprioceptive Antiedema Therapy TAPA:
  TAPA involves an intervention protocol composed of:
  * 10-min neuro dynamics oriented to the activity
  * 10-min proprioceptive neuromuscular facilitation activities.
  * 10-min proprioceptive anti-edema bandaging, including patient and/or caretaker instructions for placement, as well as assistance on techniques to use for performing everyday activities,
  Complex or combined decongestive physical therapy (CDT):
  skin care and patient education, manual lymphatic drainage MLD, joints exercises, and compression garments
  Arms: Experimental: group C:

SUMMARY:
Ninety -three female patients suffering from shoulder dysfunction after breast cancer-related arm lymphedema, will National Cancer Institute (Cairo university) be randomly distributed into three groups equal in number.

DETAILED DESCRIPTION:
In this study the patients will be randomly assigned into three groups (Thirty - one patient for each group):

Group (A):

Thirty-one patients will receive: Scapular PNF technique, Activity-Oriented Antiedema Proprioceptive Therapy (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT).

Group (B):

Thirty-one patients will receive Scapular PNF technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT))

Group (C):

Thirty-one patients will receive Activity-Oriented Antiedema Proprioceptive Therapy (TAPA) technique for the affected shoulder region plus conventional physiotherapy program in a form of (Complex decongestive therapy (CDT)

.

ELIGIBILITY:
Inclusion Criteria:

The subject selection will be according to the following criteria:

* Age range between 40-60 years.
* Only female patients will participate in the study.
* All female patients diagnosed as unilateral breast cancer.
* All Female patients operated on for BC with BCRL in stages I and II.
* All female patients suffering from shoulder dysfunction after breast cancer-related arm lymphedema.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Patients with health problems, diseases or dysfunctions that prevented them from participating in the intervention.
* Patients with bilateral lymphedema.
* Patients with previous primary lymphedema.
* Patients with metastasis.
* Patients whom staging was not possible due to atypical findings or poor image.
* Patients with active arm infection.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female patients will participate in the study
Enrollment: 93 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Cone formula for lymphedema assessment | three months
  the truncated cone formula. V = h C12 + C1C2 + C22 =12 (where V = extremity volume, h = height, C1 = circumference of the top of the cone, C2 = circumference of the base of the cone) as both extremities will be measured from the wrist to the top of the arm (axillary fold) at 4-cm intervals
Digital inclinometer for scapular range and shoulder range assessment | three months
  The digital inclinometer demonstrates moderate to excellent reliability in evaluating both shoulder and scapular range in case of shoulder disorder
Upper limb function/activity performance: Measured with e Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH): | three months
  The arm, shoulder, and hand problems quick questionnaire (Quick-Dash) used to evaluate the symptom severity and functional capacity of the patients

CONTACTS AND LOCATIONS:
Overall Officials: rasha ahmed, master, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt